CLINICAL TRIAL: NCT03622047
Title: Comparison of Epidural Labor Analgesia With Dexmedetomidine or Sufentanil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Women and children's hospital of Jiaxing university (Unknown); Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, Zeyong Yang, Department of Anesthesiology, Principal Investigator, Clinical Professor,International Peace Maternity and Child Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: International Peace Xuhui
Record Dates: First submitted 2018-07-09; First posted 2018-08-09 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Pharmacological Action
Keywords: Labor, Analgesia, Dexmedetomidine, Sufentanil
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dexmedetomidine ropivacaine (Experimental): Observing 0.5 μ g / ml dexmedetomidine + 0.1 % ropivacaine with 2 hours after fetal delivery, and the patients leave the delivery room without abnormality.
  Interventions: Drug: Dexmedetomidine ropivacaine; Drug: No analgesia labor
- sufentanil ropivacaine (Experimental): compare the analgesic effects of dexmedetomidine or sufentanil combined with ropivacaine in epidural labor.
  Interventions: Drug: Dexmedetomidine ropivacaine; Drug: No analgesia labor
- No analgesia labor (Experimental): Observing with 2 hours after fetal delivery, and the patients leave the delivery room without abnormality.
  Interventions: Drug: Dexmedetomidine ropivacaine; Drug: No analgesia labor

INTERVENTIONS:
Drug: Dexmedetomidine ropivacaine — Observing the effect of 0.5 μ g / ml sufentanil+ 0.1 % ropivacaine with 2 hours after fetal delivery, and the patients leave the delivery room without abnormality.
  Other Names: sufentanil ropivacaine
Drug: No analgesia labor — No analgesia labor control group
  Other Names: No analgesia labor control

SUMMARY:
The participants: 1800 full-term primiparas will be selected with ASA I-Ⅱgrade, 20 to 35 years old and weighing 55 to 90 kg in the investigator's hospital from may 2018 to December 2018. 1200 primiparas were divided into A and B according to the computer randomized numbers, and 600 parturients without labor analgesia in the same period were selected as group C, with 600 patients in each group. All parturients signed the informed consent form and were approved by the hospital ethics Committee.

DETAILED DESCRIPTION:
1200 primiparas were divided into A and B according to the computer randomized numbers, and 600 parturients without labor analgesia in the same period were selected as group C, with 600 patients in each group. All parturients signed the informed consent form and were approved by the hospital ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-Ⅱ, aged 22 - 42,
* gestational age ≥ 37, weight 55 - 90 kg,
* labor analgesia is required by full-term primiparas.

Exclusion Criteria:

* serious cardiovascular and cerebrovascular system diseases,
* bradycardia, conduction block
* fetal distress
* contraindications of intraspinal anesthesia.

Ages: 22 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 1800 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
The onset time | 30 minutes
  A drug's effects to come to prominence upon administration.

SECONDARY OUTCOMES:
analgesic effect | 1 day
  VAS Score Visual analogue scale (VAS) of pain before and after analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Yongtao Gao, MD, Study Director — Shanghai Jiao Tong University School of Medicine
Locations (1):
- International Peace Maternity and Child Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No